CLINICAL TRIAL: NCT04697381
Title: A PHASE 3 MULTICENTER, OPEN LABEL, MULTI COHORT STUDY TO EVALUATE THE EFFICACY AND SAFETY OF SOMATROPIN IN JAPANESE PARTICIPANTS WITH PRADER-WILLI SYNDROME (PWS)
Brief Title: Study of the Efficacy and Safety of Somatropin in Japanese Participants With PWS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6281323; 2024-000101-32 (Registry Identifier: EudraCT); NCT04697381 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- somatropin - GH naïve pediatric cohort (Experimental): All participants will receive somatropin.
  Interventions: Biological: somatropin - GH naïve pediatric cohort
- somatropin - GH treated pediatric cohort (Experimental): All participants will receive somatropin
  Interventions: Biological: somatropin - GH treated cohort
- somatropin - adult cohort (Experimental): All participants will receive somatropin
  Interventions: Biological: somatropin - adult cohort

INTERVENTIONS:
Biological: somatropin - GH naïve pediatric cohort — somatropin 0.245 mg/kg/week
  Arms: somatropin - GH naïve pediatric cohort
Biological: somatropin - GH treated cohort — somatropin 0.084 mg/kg/week
  Arms: somatropin - GH treated pediatric cohort
Biological: somatropin - adult cohort — somatropin 0.084 mg/kg/week
  Arms: somatropin - adult cohort

SUMMARY:
This is a multicenter, open label, multi cohort study to evaluate the efficacy and safety of somatropin in a cohort of Japanese participants with PWS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with documentation of genetically confirmed diagnosis of PWS.
2. No plan to initiate a new treatment that may affect the body composition, such as gonadal hormone replacement therapy.
3. Currently on appropriate diet and exercise programs and willing to continue throughout the study period at the discretion of the investigator.
4. Participants, and if required by local/site regulations their parent(s)/legal guardian(s) must be willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
5. Evidence of a personally signed and dated ICD (and written assent where applicable based on age and country regulation) indicating that the participant or a legally acceptable representative/parent(s)/legal guardian has been informed of all pertinent aspects of the study. Refer to Appendix 1 for the detailed process of obtaining consent.

   For inclusion of GH naïve pediatric cohort, participants must meet criteria 6 to 8:
6. 18 years or younger.
7. Naïve to GH treatment.
8. Tanner stage 1 (for testes in males, for breasts in females).

   For inclusion of GH treated pediatric cohort, participants must meet criteria 9 and 10:
9. Continued GH treatment for at least 2 years with stable dose for the last 6 months and being on GH at time of inclusion. The recent dose should be higher than 0.084 mg/kg/week.
10. Participants who are about to complete GH treatment for his/her short stature (eg, due to meeting the treatment stopping criteria defined as a height SDS more than -2.5 for Japanese adult standards).

    For inclusion of adult cohort, participants must meet criteria 11 to 13:
11. 18 years of chronological age or older at Day 1 visit.
12. Off from GH treatment for at least 1 year.
13. Serum IGF-I level within +2 SDS, adjusted for age and sex.

Exclusion Criteria:

1. Participants with uncontrolled diabetes at the discretion of the investigator.
2. Participants with malignant tumors.
3. Participants with severe obesity or serious respiratory impairment.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half- lives preceding the first dose of study intervention used in this study (whichever is longer).
6. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Japan (5):
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Osaka Women's and Children's Hospital, Izumi, Osaka
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - National Center for Child Health and Development, Setagaya-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kawai M, Murakami N, Horikawa R, Muroya K, Fujisawa Y, Hoshino Y, Okayama A, Sato T, Ebata N, Ogata T. Improvement in body composition of Japanese participants with Prader-Willi syndrome following somatropin treatment: an open-label, multi cohort Phase 3 study. Endocr J. 2025 Aug 1;72(8):925-935. doi: 10.1507/endocrj.EJ24-0659. Epub 2025 May 28. PMID 40436776
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6281323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with Prader-Willi syndrome (PWS ) received somatropin, a recombinant human growth hormone (r-hGH) in this study.
Pre-assignment Details: This study had 3 cohorts (GH naive pediatric cohort, GH treated pediatric cohort and adult cohort).
Groups:
- GH Naive Pediatric Cohort: Participants 18 years or younger, naive to GH treatment, received somatropin 0.245 milligram per kilogram per week (mg/kg/week) subcutaneously. Treatment period was of 12 months and extension period was of 36 months. Participants were followed up to 28 days.
- GH Treated Pediatric Cohort: Participants 18 years or younger, who continued GH treatment for at least 2 years with stable dose for the last 6 months and were on GH at time of inclusion, received somatropin 0.084 mg/kg/week subcutaneously. The dosage was adjusted according to participants symptoms and insulin-like growth factor 1 (IGF-1) levels with maximum dose up to 1.6 mg/day. Treatment period was of 12 months and extension period was of 36 months. Participants were followed up to 28 days.
- Adult Cohort: Adult participants who were off from GH treatment for at least 1 year, initially received somatropin 0.042 mg/kg/week subcutaneously. Dose was titrated up to 0.084 mg/kg/week from Month 1 visit. The dosage was adjusted according to participants symptoms and serum IGF-1 levels with maximum dose up to 1.6 mg/day. Treatment period was of 12 months and extension period was of 36 months. Participants were followed up to 28 days.
Period: Treatment Period
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort | Adult Cohort
Started | 6 | 7 | 20
Completed | 6 | 7 | 20
Not Completed | 0 | 0 | 0
Period: Extension Period
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort | Adult Cohort
Started | 6 | 7 | 20
Completed | 6 | 7 | 14
Not Completed | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GH Naive Pediatric Cohort: Participants 18 years or younger, naive to GH treatment, received somatropin 0.245 mg/kg/week subcutaneously. Treatment period was of 12 months and extension period was of 36 months. Participants were followed up to 28 days.
- GH Treated Pediatric Cohort: Participants 18 years or younger, who continued GH treatment for at least 2 years with stable dose for the last 6 months and were on GH at time of inclusion, received somatropin 0.084 mg/kg/week subcutaneously. The dosage was adjusted according to participants symptoms and IGF-1 levels with maximum dose up to 1.6 mg/day. Treatment period was of 12 months and extension period was of 36 months. Participants were followed up to 28 days.
- Total: Total of all reporting groups
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort | Adult Cohort | Total
Number analyzed (Participants) | 6 | 7 | 20 | 33
Age, Customized [Count of Participants; unit: Participants]
  Less than (<6) years | 3 | 0 | 0 | 3
  6-12 years | 3 | 1 | 0 | 4
  13-17 years | 0 | 5 | 0 | 5
  18-44 years | 0 | 1 | 20 | 21
  More than equal to (>=) 45 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 13 | 18
  Male | 4 | 4 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 20 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 7 | 20 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 12 in Lean Body Mass Measured by Dual-Energy X-ray Absorptiometry (DEXA): Adult Cohort
Description: Lean body mass, a measurement of body composition, was assessed by DEXA scan, and calculated as lean body mass (%) = lean body mass kilogram (kg) / (lean body mass [kg] + fat mass [kg]) *100.
Time Frame: Baseline, Month 12
Population: Efficacy evaluable set included all participants assigned to study intervention and who took at least one dose of study intervention and had at least one efficacy evaluation. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and this time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of body mass
Arm/Group | Adult Cohort
Number analyzed (Participants) | 19
Percentage of body mass | 3.09 [1.85 to 4.33]

2. Primary Outcome: Change From Baseline to Month 12 in Lean Body Mass Measured by DEXA: GH Naive Pediatric and GH Treated Pediatric Cohort
Description: Lean body mass, a measurement of body composition, was assessed by DEXA scan, and calculated as lean body mass (%) = lean body mass (kg) / (lean body mass [kg] + fat mass [kg])*100.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of body mass
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort
Number analyzed (Participants) | 6 | 6
Percentage of body mass | 4.59 (4.490) | -1.34 (3.238)

3. Secondary Outcome: Change From Baseline to Month 12 in Lean Body Mass Measured by Bioelectrical Impedance Analysis (BIA)-Adult Cohort
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of body mass
Arm/Group | Adult Cohort
Number analyzed (Participants) | 19
Percentage of body mass | 2.03 [-0.67 to 4.73]

4. Secondary Outcome: Change From Baseline to Month 12 in Lean Body Mass Measured by BIA-GH Naive Pediatric and GH Treated Pediatric Cohort
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of body mass
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort
Number analyzed (Participants) | 6 | 5
Percentage of body mass | 3.32 (3.867) | 0.58 (4.711)

5. Secondary Outcome: Change From Baseline to Month 12 in Body Fat (Percentage) Measured by DEXA: Adult Cohort
Description: Body fat was assessed by DEXA scan. and calculated as body fat (%) = body fat (kg) / [lean body mass (kg) + body fat (kg)]*100.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of body fat
Arm/Group | Adult Cohort
Number analyzed (Participants) | 19
Percentage of body fat | -3.09 [-4.33 to -1.85]

6. Secondary Outcome: Change From Baseline to Month 12 in Body Fat (Percentage) Measured by DEXA: GH Naive Pediatric and GH Treated Pediatric Cohort
Description: as for outcome 5
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of body fat
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort
Number analyzed (Participants) | 6 | 6
Percentage of body fat | -4.59 (4.490) | 1.34 (3.238)

7. Secondary Outcome: Change From Baseline to Month 12 in Adipose Tissue Distribution Measured by Abdominal Computed Tomography (CT)
Description: Adipose tissue distribution was measured by abdominal CT. Areas of subcutaneous adipose tissue (SAT) (centimeter square [cm^2]), visceral adipose tissue (VAT) (cm^2) were measured at the level of the umbilicus by abdominal CT.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeter square (cm^2)
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort | Adult Cohort
Number analyzed (Participants) | 6 | 6 | 19
Centimeter square (cm^2)
  Change at Month 12, SAT | 60.423 (138.2001) | 102.222 (211.9111) | -13.764 (31.0212)
  Change at Month 12, VAT | 4.825 (13.5401) | -13.403 (28.5490) | -4.040 (16.8243)

8. Secondary Outcome: Change From Baseline to Month 6 in Lean Body Mass Measured by DEXA: Adult Cohort Only
Description: as for outcome 2
Time Frame: Baseline, Month 6
Population: Efficacy evaluable set included all participants assigned to study intervention and who took at least one dose of study intervention and had at least one efficacy evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of body mass
Arm/Group | Adult Cohort
Number analyzed (Participants) | 20
Percentage of body mass | 2.38 [1.30 to 3.46]

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An adverse event was any untoward medical occurrence in administered medicinal product, event need not necessarily have a causal relationship with product treatment or usage. A serious adverse event was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. Treatment emergent AEs were events emerged during treatment period and were absent before treatment or that worsened relative to pretreatment state. TEAEs consist of SAEs and non-SAEs
Time Frame: From day 1 up to 28 days after end of study treatment (maximum duration up to 38 months)
Population: Full analysis set (FAS) included all participants assigned to study intervention and who took at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort | Adult Cohort
Number analyzed (Participants) | 6 | 7 | 20
Participants
  TEAEs | 5 | 7 | 19
  Treatment Emergent SAEs | 0 | 1 | 3

10. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for abnormal laboratory values for chemistry parameters: alanine aminotransferase, alkaline phosphatase greater than (>) 3.0*upper limit of normal (ULN), albumin > 1.2*ULN, urea nitrogen millimoles per liter (mmol/L) > 1.3*ULN, HDL cholesterol mmol/L less than (<) 0.8* lower limit of normal (LLN), LDL cholesterol mmol/L >1.2*ULN, triglycerides mmol/L > 1.3*ULN, thyrotropin milliunits per liter (mU/L) <0.8*LLN and >1.2*ULN, glucose (mmol/L) >1.5*ULN, hemoglobin A1C liter of cells per liter of blood (L/L) >1.3*ULN.
Time Frame: From Day 1 up to 28 days after end of study treatment (maximum duration up to 38 months)
Population: FAS included all participants assigned to study intervention and who took at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort | Adult Cohort
Number analyzed (Participants) | 6 | 7 | 20
Participants | 5 | 3 | 16

11. Secondary Outcome: Bone Maturation
Description: Bone maturation is the process whereby the tissue undergoes changes from the embryonic rudiment of bone to the adult form. Bone maturation was calculated as bone age divided by chronological age. Participants with bone maturation value greater than 1 is presented in this outcome measure.
Time Frame: 12 months
Population: FAS included all participants assigned to study intervention and who took at least one dose of study intervention.
Measure: Number; unit: Participants
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort
Number analyzed (Participants) | 6 | 7
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to 28 days after end of study treatment (maximum duration up to 38 months)
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Analysis population include all participants assigned to study intervention and who took at least one dose of study intervention.
Arm/Group | GH Naive Pediatric Cohort | GH Treated Pediatric Cohort | Adult Cohort
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7 | 3/20
Other Adverse Events (participants affected / at risk) | 5/6 | 7/7 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GH Naive Pediatric Cohort (N=6) | GH Treated Pediatric Cohort (N=7) | Adult Cohort (N=20)
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GH Naive Pediatric Cohort (N=6) | GH Treated Pediatric Cohort (N=7) | Adult Cohort (N=20)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Anal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Extravasation (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 3 | 1 | 11
Cellulitis (Infections and infestations) | 0 | 0 | 1
Eczema impetiginous (Infections and infestations) | 0 | 0 | 2
Genital candidiasis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 2
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 4
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 3
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 1
Body height increased (Investigations) | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 3
Insulin-like growth factor increased (Investigations) | 1 | 1 | 3
Liver function test increased (Investigations) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 1 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Pseudohypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1
Dissociative disorder (Psychiatric disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1
Eczema eyelids (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Hypoaesthesia teeth (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Genital abscess (Infections and infestations) | 0 | 0 | 1
Herpangina (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Genital tract inflammation (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2
Dysphoria (Psychiatric disorders) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT04697381/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT04697381/SAP_001.pdf